CLINICAL TRIAL: NCT00375960
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Crossover Study of the Safety, Efficacy and Pharmacokinetics of Two Escalating, Oral Doses of V3381 (200 mg BID and 400 mg BID) for 28 Days in Patients With Diabetic Peripheral Neuropathic Pain (DPNP)
Brief Title: A Research Study of V3381 for the Treatment of Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vernalis (R&D) Ltd (Industry)
Collaborators: Cita NeuroPharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: V3381-2DPNP01
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2007-04-02 (Estimated); Status verified 2007-03

CONDITIONS: Pain; Diabetic Neuropathies
Keywords: Pain associated with diabetes Type I or Type II; Neuropathic Pain due to diabetes; Diabetic peripheral neuropathic pain; Pain; Diabetes with burning sensation in the arms and/or legs; Diabetes with tingling sensation in the arms and/or legs; Neuropathic Pain Due to Diabetes Type I or Type II
MeSH Terms: conditions — Pain; Diabetic Neuropathies

INTERVENTIONS:
Drug: V3381
Drug: Placebo

SUMMARY:
The objective of this study is to investigate the safety and efficacy of an investigational drug, V3381, for the treatment of diabetic peripheral neuropathic (DPN) pain (pain in one's feet and legs, or even in one's hands and arms, sometimes experienced by people with diabetes). An investigational drug is one that is not approved by the United States Food and Drug Administration (FDA) and/or Health Canada.

DETAILED DESCRIPTION:
Diabetic Peripheral Neuropathic Pain (DPNP) is pain in your feet and legs, or even in your hands and arms, sometimes experienced by people with diabetes. Neuropathic pain syndromes are much more common than is perhaps generally recognized. Approximately 1% of the population in western countries suffers from neuropathic pain. Some clinical conditions are associated with a relatively high incidence of neuropathic pain. Approximately 15% of patients with diabetic neuropathy have persistent neuropathic pain in the feet, legs and hands.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18-75 years of age
* Diabetes mellitus (type I or type II)
* No change in medications for reducing blood sugar within 4 weeks before screening
* Experiencing daily pain due to diabetic neuropathy for at least 6 months but not more than 5 years
* Neuropathic pain must begin in the feet, with relatively symmetrical onset.
* Willing to perform self-monitoring of blood glucose
* Able to communicate intelligibly with the investigator and study coordinator
* Keeping all appointments for clinic visits, tests, and procedures

Exclusion Criteria:

* Any clinically significant neurologic disorders (with the exception of diabetic peripheral neuropathic pain)
* Any clinically significant or unstable medical or psychiatric condition that would interfere with the patient's ability to participate in the study
* Prior renal transplant or current renal dialysis
* Pernicious anemia
* Untreated hypothyroidism
* Amputations due to diabetes mellitus (with the exception of toes)
* Any clinically significant abnormal electrocardiogram (ECG)
* Any history of cardiac arrhythmia
* History of myocardial infarction
* Active angina
* Uncontrolled hypertension (i.e., > 140/90 mm Hg)
* Known or at high risk of hepatitis B or C infection
* Known or at high risk of human immunodeficiency virus (HIV) infection
* Any anticipated need for surgery during the study
* Glycosylated hemoglobin (HbA1c) > 9%
* Known seizure disorder
* Any malignancy in the past 2 years (with the exception of basal cell carcinoma)
* Pain that cannot be clearly differentiated from, or conditions that interfere with the assessment of diabetic neuropathic pain.
* Use of anticonvulsants, antidepressants, or prescription membrane-stabilizing agents
* History of substance abuse or dependence within the past year, excluding nicotine and caffeine
* Frequent and/or severe allergic reactions with multiple medications
* Participation in any clinical trial within 30 days before screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-06; Study Completion 2007-04

PRIMARY OUTCOMES:
11 point numerical pain rating scale (NPRS) daily diary

SECONDARY OUTCOMES:
Modified Brief Pain Inventory for DPN
McGill Pain Questionnaire - Short Form
Neuropathic Pain Symptom Inventory
Medical Outcomes Survey Short Form - 12, Version 2
Patient Global Impression of Change
Patient Preference Questionnaire (end of 2nd treatment period only)
Clinical Global Impression of Change
Additional secondary assessments will be included in the daily diary: consumption of rescue analgesics
daily sleep interference score

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sang, M.D., MPH, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (6):
- United States (5):
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Translational Pain Research Group, Brigham & Women's Hospital, Boston, Massachusetts
  - American Center for Clinical Trials, Southfield, Michigan
  - Diabetes & Glandular Disease Research Associates Inc., San Antonio, Texas
- LMC Endocrinology Centres Ltd., Thornhill, Ontario, Canada